CLINICAL TRIAL: NCT03601403
Title: Tablet-assisted Training as a Complement Hospital Intervention in Patients With Acute Exacerbations of COPD
Brief Title: Tablet-assisted Training in Exacerbated COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DF0075UG
Record Dates: First submitted 2018-07-04; First posted 2018-07-26 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Education; Dry Powder Inhalers; Metered Dose Inhalers; Pulmonary Disease; Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (No Intervention): Received the standard medical and pharmacological care provided by the hospital
- Inhaler technique (Experimental): The intervention group received the standard medical and pharmacological care provided by the hospital. In addition, a tablet-assisted training on the use of inhalers, which included an explanation of the use of inhalers together with a ventilatory re-education program.
  Interventions: Device: inhaler technique

INTERVENTIONS:
Device: inhaler technique — The first day of the intervention consisted primarily of ventilatory re-education. During the realization of the technique, he was videotaped with a Tablet so that later the patient could be seen and on the video to be able to give him the guidelines for the correction. On the second and third day of the intervention, ventilation re-education was performed and the inhalation technique was subsequently trained.
  Arms: Inhaler technique

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a public health problem with great morbidity. The main therapeutic strategy is inhalers. The objective of this study is to determine the efficacy of a tablet-assisted training in the use of inhalers in patients with COPD including ventilatory re-education and video recordings of the patients themselves.

DETAILED DESCRIPTION:
The importance of this pathology lies not only in its high prevalence, which is expected to increase due to the aging of society but also in its high mortality. In Europe, it is estimated that 50% of adult patients do not use the inhaler correctly. The clinical development of COPD includes periods of stability interspersed with symptomatic exacerbations, which usually involve hospitalization. During these hospitalizations, respiratory symptoms are worsening.Nevertheless, in Europe, it is estimated that 50% of adult patients do not use the inhaler correctly. Thus, it is very important the pharmacological education in this patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of exacerbation of COPD.
* To possess pharmacological treatment in the form of inhalers.

Exclusion Criteria:

* Inability to provide informed consent.
* Presence of psychiatric or cognitive disorders.
* Organ failure or cancer.
* Inability to cooperate.
* Patients who had experienced an exacerbation in the last month.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-06-23 (Actual); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in the first second (FEV1) | [Time Frame: baseline, 12 months]
  Changes from baseline to postintervention in FEV1vas evaluated by a spirometer.

SECONDARY OUTCOMES:
Knowledge of the Chronic Obstructive Pulmonary Disease | [Time Frame: Baseline, 12 months]
  Evaluated at baseline by Chronic Obstructive Pulmonary Disease Questionnaire (COPD-Q). COPD knowledge was evaluated using the Chronic Obstructive Pulmonary Disease Knowledge Questionnaire (COPD-Q; Maples, Franks, Ray, Stevens, & Wallace, 2010). The COPD-Q is a valid, readable, and reliable 13-item (each one score 0 to 3) self-administered true/false questionnaire assessing COPD knowledge in patients with low health literacy skills. A higher punctuation indicates better results.
Cognitive Level | [Time Frame: Baseline]
  Cognitive level was assessed using the Montreal Cognitive Assessment (MOCA).
Functional independence | [Time Frame: Baseline]
  Functional independence was assessed using the Functional Independence Mease Scale (FIM). This scale has 18 items that are grouped into 2 dimensions, 13 motor items, and 5 cognitive items. The total score range between 18 points (total dependence) to 126 points (Independence completes).
Anxiety-depression level | [Time Frame: Baseline, 12 months]
  Changes from baseline to postintervention in anxiety and depression measured with the Hospital Anxiety and Depression Scale. Patients are going to complete this questionnaire composed of statements relevant to either generalized anxiety or depression. It is composed of 14 items, 7 for anxiety and 7 for depression and higher values are related to higher depression and anxiety.
Adhesion to inhalers | [Time Frame: Baseline]
  Level of adhesion to inhalers was assessed with TAI (Inhaler Adhesion Test).
Dyspnea level | [Time Frame: Baseline]
  Perceived perception of dyspnea was collected through the Modified Borg Scale. Patients have to choose a number between 0 ( no dyspnea) to 10 (higher dyspnea).
Physical fitness | [Time Frame: baseline, 12 months]
  Physical fitness was assessed by performing the five-times-sit-to-stand test. It consists of getting up and sitting five times in a row without a support. The time period in which the exercise is performed is the patient's score with a maximum of 60 seconds
Technique of the inhaler | [Time Frame: baseline, 12 months]
  The evaluation of the technique of the inhalers was carried out by means of a checklist composed of 5 items. Checked those points that were done correctly obtaining 5 points if the technique that was done correctly.
Pressure expiratory force (PEF) | [Time Frame: baseline, 12 months]
  Changes from baseline to postintervention in PEF were assessed using a peak flow.

CONTACTS AND LOCATIONS:
Overall Officials: M. Carmen Valenza, PH MD, Principal Investigator — Department of Physical Therapy. University of Granada.
Locations (1):
- Faculty of Health Sciences. University of Granada., Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided